CLINICAL TRIAL: NCT06389240
Title: Early Weight Bearing in Unicondylar Tibial Plateau Fractures: How Does it Affect Gait Pattern, Mobility and Overall Outcome: A Randomized Controlled Trial
Brief Title: Early Weight Bearing in Unicondylar Tibial Plateau Fractures
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Justin Haller, Principle Investigator, University of Utah
Other Study IDs: 160848
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Early Mobilization
Keywords: unicondylar tibia plateau fractures; early mobilization; Gait analysis
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- 6 weeks post-operatively early weight bearing: Full weight bearing will be allowed 6 weeks post-operatively. Gait analyses is carried out on when full weight-bearing is allowed.
  Interventions: Other: 6 weeks post-operatively early weight bearing
- 10 weeks post-operatively weight bearing (standard of care): Full weight bearing will be allowed 10 weeks post-operatively. Gait analyses is carried out on when full weight-bearing is allowed.
  Interventions: Other: 10 weeks post-operatively weight bearing (standard of care)

INTERVENTIONS:
Other: 6 weeks post-operatively early weight bearing — Early mobilization 6 weeks post-operatively. Gait analyses is carried out on when full mobilization is allowed. Gait analysis is performed while using force-measuring insoles (loadsol, Novel).
  Groups: 6 weeks post-operatively early weight bearing
Other: 10 weeks post-operatively weight bearing (standard of care) — Standard of care mobilization at 10 weeks post-operatively. Gait analyses is carried out on when full mobilization is allowed. Gait analysis is performed while using force-measuring insoles (loadsol, Novel).
  Groups: 10 weeks post-operatively weight bearing (standard of care)

SUMMARY:
The investigators aim of the study is to assess the effects of early mobilization after surgically treated unicondylar tibia plateau fractures (6 weeks without weight bearing) on gait, patient satisfaction, return to work/sports and complication rate. The data will be compared to a 10-12 week non-weight bearing group (standard of care).

It is assumed that earlier mobilization does not lead to an increase in the complications - in particular osteosynthesis failure and infections -, but leads to improved patient satisfaction, reduced return to work/sports times, and has a positive impact on the overall outcome

DETAILED DESCRIPTION:
Tibial plateau fractures are common sports injuries caused by accidents such as skiing and mountain biking. Thus, young adults with high functional and athletic demands are often affected. The best possible restoration of the original joint function and resilience is therefore particularly important for this group of patients. In addition, prolonged immobilization in this patient group poses a high risk of loss of earnings and a significant impairment in athletic performance.

These injuries usually require surgical treatment which is followed by 10-12 weeks without weight bearing. In recent years, there has been a shift towards earlier mobilization with many injuries. In addition, numerous studies showed the negative effects of prolonged immobility. Nevertheless, these negative effects must always be weighed against the possibility of osteosynthesis failure.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, at least 18 years of age, max 65 years of age
* Unilateral tibial plateau fracture AO:41b/c
* Written consent to participate (consent can be revoked at any time without giving reasons)
* Surgery during the study period
* Follow-up on-site (Salt Lake City, Utah, United States)

Exclusion Criteria:

* Multiple injured or polytraumatized patients
* Other injuries or illnesses that impair the patient's mobility or gait
* Cognitive limitations such as dementia, delirium or similar disease
* Refusal to participate
* Severe underlying disease with significant limitations in the ability to regenerate e.g.

malignancies

* Pathologic or osteoporotic fractures
* Unable to attend clinic in person for follow-ups
* pregnant women and fetus

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients,18 - 65 years of age with a unilateral tibial plateau fracture.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-12-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Average peak load (Newtons (N)) | 6 weeks for early mobilization group
  Gait analysis is performed while using force-measuring insoles. Patients are asked to complete an parcours with the force-measuring insoles (stand up from a chair with armrests, walk 10 meters, turn, walk back and sit down again. Afterwards (if possible), 5 steps with a handrail should be climbed up and down.
Average peak load (Newtons (N)) | 10 weeks for standard of care (SOC) group
  Gait analysis is performed while using force-measuring insoles. Patients are asked to complete an parcours with the force-measuring insoles (stand up from a chair with armrests, walk 10 meters, turn, walk back and sit down again. Afterwards (if possible), 5 steps with a handrail should be climbed up and down.
Average peak load (Newtons (N)) | 1 week after full weight bearing is allowed for both 6 week early mobilization and SOC groups.
  Gait analysis is performed while using force-measuring insoles. Patients are asked to complete an parcours with the force-measuring insoles (stand up from a chair with armrests, walk 10 meters, turn, walk back and sit down again. Afterwards (if possible), 5 steps with a handrail should be climbed up and down.
Average peak load (Newtons (N)) | 2 weeks after full weight bearing is allowed for both 6 week early mobilization and SOC groups.
  Gait analysis is performed while using force-measuring insoles. Patients are asked to complete an parcours with the force-measuring insoles (stand up from a chair with armrests, walk 10 meters, turn, walk back and sit down again. Afterwards (if possible), 5 steps with a handrail should be climbed up and down.
Average peak load (Newtons (N)) | 6 weeks after full weight bearing is allowed for both 6 week early mobilization and SOC groups.
  Gait analysis is performed while using force-measuring insoles. Patients are asked to complete an parcours with the force-measuring insoles (stand up from a chair with armrests, walk 10 meters, turn, walk back and sit down again. Afterwards (if possible), 5 steps with a handrail should be climbed up and down.
Average peak load (Newtons (N)) | 12 weeks after full weight bearing is allowed for both 6 week early mobilization and SOC groups.
  Gait analysis is performed while using force-measuring insoles. Patients are asked to complete an parcours with the force-measuring insoles (stand up from a chair with armrests, walk 10 meters, turn, walk back and sit down again. Afterwards (if possible), 5 steps with a handrail should be climbed up and down.
Average peak load (Newtons (N)) | 6 months after full weight bearing is allowed for both 6 week early mobilization and SOC groups.
  Gait analysis is performed while using force-measuring insoles. Patients are asked to complete an parcours with the force-measuring insoles (stand up from a chair with armrests, walk 10 meters, turn, walk back and sit down again. Afterwards (if possible), 5 steps with a handrail should be climbed up and down.

CONTACTS AND LOCATIONS:
Overall Officials: Justin Haller, M.D., Principal Investigator — University of Utah Orthopaedics
Locations (1):
- University of Utah Orthopedics, Salt Lake City, Utah, United States